CLINICAL TRIAL: NCT07337187
Title: The Effect of Thread-Embedding Acupuncture at EX-B2 Acupoint on Pain Intensity and Quality of Life in Patients With Chronic Low Back Pain
Brief Title: Effect of Thread-Embedding Acupuncture at EX-B2 on Pain and Quality of Life in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Atalya Vetta Widarto, MD, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 25111755
Record Dates: First submitted 2025-12-18; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Low Back Pain
Keywords: Chronic Low Back Pain; Lumbago
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Thread-embedding acupuncture and analgesic therapy will be designated as the intervention group, while sham thread-embedding acupuncture and analgesic therapy will be designated as the control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: the participants and the outcome assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thread-embedding acupuncture (Experimental): Thread-embedding acupuncture and analgesic therapy
  Interventions: Device: Thread-embedding acupuncture
- Sham thread-embedding acupuncture (Sham Comparator): Sham thread-embedding acupuncture and analgesic therapy
  Interventions: Device: Sham Thread-embedding acupuncture

INTERVENTIONS:
Device: Thread-embedding acupuncture — Thread-embedding acupuncture is performed bilaterally at a pair of lumbar EX-B2 points using needles containing polydioxanone (PDO) threads, positioned 12.5 mm lateral to the spinous processes. The targeted EX-B2 level is selected from L1 to L5 based on the subject's main pain location, informed by dermatome and myotome mapping and lumbar segmental concepts.
  Arms: Thread-embedding acupuncture
Device: Sham Thread-embedding acupuncture — Sham thread-embedding acupuncture is performed bilaterally at the lumbar EX-B2 points using needles that are placed in contact with the skin at the acupuncture point sites without skin penetration. The targeted EX-B2 level is selected from L1 to L5 based on the subject's predominant pain location, guided by dermatome and myotome mapping and the principles of lumbar segmental innervation.
  Arms: Sham thread-embedding acupuncture

SUMMARY:
The goal of this clinical trial is to learn whether thread-embedding acupuncture (TEA) is more effective than sham thread-embedding acupuncture in treating adults with chronic low back pain. The study will also evaluate the safety of TEA.

The main questions it aims to answer are:

* Does TEA reduce pain intensity more effectively than sham TEA?
* Does TEA improve quality of life compared with sham TEA?
* Does TEA reduce the frequency of bothersome pain episodes?
* Does TEA reduce the use of routine and additional (extra) pain medications?
* What side effects occur in participants receiving TEA compared with sham TEA?

Researchers will compare TEA with sham TEA (a procedure that mimics acupuncture without needle insertion or thread placement) to determine whether TEA provides greater and longer-lasting benefits for chronic low back pain.

Participants will:

* Receive a single session of TEA or sham TEA
* Continue using pain medications as prescribed by their physician
* Be evaluated at weeks 2, 4, 6, and 8 after treatment
* Complete pain assessments, quality-of-life questionnaires, and reports of pain episodes and medication use
* Attend in-person clinic visits at weeks 4 and 8, and receive telephone follow-ups at weeks 2 and 6

DETAILED DESCRIPTION:
* In the intervention group, thread-embedding acupuncture is performed using needles containing polydioxanone (PDO) threads at the bilateral lumbar EX-B2 acupuncture points (12.5 mm lateral to the spinous process).
* In the control group, the needle is only touched to the skin at the acupuncture point area without skin penetration.
* The selection of the EX-B2 level is based on the vertebral segment from L1 to L5 that best corresponds to the subject's dominant pain location, with reference to dermatome and myotome mapping as well as the concept of lumbar segmental innervation. If available, supporting examination results (e.g., MRI or CT scan) indicating abnormalities at a specific segment are used as additional references. When more than one segment is considered possible, the midpoint level is selected.
* After completion of the study, participants in the sham thread-embedding acupuncture group are allowed to receive actual thread-embedding acupuncture therapy for chronic low back pain.

Outcome Definitions

- Bothersome pain episodes: The number of days in the past 7 days during which the subject experienced bothersome low back pain.

Bothersome low back pain is defined as pain that is sufficiently significant to interfere with daily activities, rest, concentration, or overall comfort. Mild pain or pain that does not interfere with activities is not counted.

- Frequency of routine analgesic use: The number of days in the past 7 days during which the subject consumed routine analgesic medication (taken as prescribed by a physician).

Routine analgesics may include primary analgesics (paracetamol and/or opioids) and/or adjuvant analgesics (muscle relaxants, antiepileptics, antidepressants, antispasmodics).

- Frequency of additional (rescue) analgesic use: The number of days in the past 7 days during which the subject consumed additional (as-needed) analgesic medication when pain remained bothersome.

Additional analgesics may include primary analgesics (paracetamol and/or opioids) and/or adjuvant analgesics (muscle relaxants, antiepileptics, antidepressants, antispasmodics).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥18 years
* Subjects with low back pain lasting for at least 3 months (>12 weeks)
* Maximum low back pain intensity within the past 2 weeks of ≥3 on a 0-10 scale, measured using the Numeric Pain Rating Scale (NPRS) or the Face, Legs, Activity, Cry, Consolability (FLACC) scale
* Willing to participate in the study until completion and able to provide written informed consent
* Receiving pharmacological therapy with a stable analgesic regimen for at least the past 2 weeks, which may include non-opioid analgesics (paracetamol), opioid analgesics (codeine, tramadol, morphine), antidepressants (amitriptyline, duloxetine), anticonvulsants (gabapentin, pregabalin, carbamazepine), and/or muscle relaxants (eperisone, baclofen)

Exclusion Criteria:

* History of hypersensitivity to acupuncture or thread-embedding acupuncture (TEA), including allergy to stainless steel or polydioxanone threads
* History of keloid formation or skin disorders at the planned TEA insertion sites in the low back area
* Presence of specific spinal pathology, including fracture, tumor, infection, or severe lumbar spinal stenosis (Schizas grade C or D) requiring surgical intervention
* Structural spinal abnormalities (scoliosis or kyphosis) detected on physical examination
* History of spinal surgery or current indication for spinal surgery due to severe neurological deficits
* Presence of other chronic pain syndromes (fibromyalgia, myofascial pain syndrome, neuropathic pain syndrome, arthritis, chronic pelvic pain, migraine, or chronic tension-type headache) or severe comorbidities (stroke with sensory deficits, Parkinson's disease, end-stage chronic kidney disease, or terminal heart failure) that may affect pain assessment
* Presence of cardiac disease, hematologic disorders, or uncontrolled diabetes mellitus
* Regular use of systemic steroids, nonsteroidal anti-inflammatory drugs (NSAIDs), antiplatelet agents, anticoagulants, or topical analgesics
* Body mass index (BMI) <18 kg/m²
* Receive other therapies for low back pain, including dry needling, neuromuscular taping, or acupuncture within the past 2 weeks, or thread-embedding acupuncture within the past 6 months
* Receive spinal interventional therapy (surgery or injection) within the past 3 months, or stem cell therapy for chronic low back pain within the past 12 months
* Cognitive impairment or other neurological disorders, severe psychiatric or psychological conditions, or a history of alcohol or substance abuse
* Pregnant or breastfeeding women, or women planning to become pregnant within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Before therapy, week 2, week 4, week 6, week 8
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS). NPRS is an 11-point numeric scale ranging from 0 to 10, where 0 = no pain and 10 = the worst pain imaginable. Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Health-Related Quality of Life | Before therapy (baseline), week 4, and week 8.
  Health-related quality of life will be assessed using the European Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire, a standardized and validated instrument.
  The EQ-5D-5L evaluates five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with five levels of severity.
  EQ-5D-5L Index Value:
  The index score is derived from the five dimensions and typically ranges from less than 0 (health states worse than death) to 1.0 (full health), with higher scores indicating better health-related quality of life.
Frequency of Bothersome Pain Episodes | Before therapy, week 2, week 4, week 6, week 8
  The number of days in the past 7 days during which the subject experienced bothersome low back pain.
  Bothersome low back pain is defined as pain that is sufficiently significant to interfere with daily activities, rest, concentration, or overall comfort. Mild pain or pain that does not interfere with activities is not counted.
Frequency of Routine Analgesic Use | Before therapy, week 2, week 4, week 6, week 8
  The number of days in the past 7 days during which the subject consumed routine analgesic medication (taken as prescribed by a physician).
  Routine analgesics may include primary analgesics (paracetamol and/or opioids) and/or adjuvant analgesics (muscle relaxants, antiepileptics, antidepressants, antispasmodics).
Frequency of Additional (extra) Analgesic Use | Before therapy, week 2, week 4, week 6, week 8
  The number of days in the past 7 days during which the subject consumed additional (as-needed) analgesic medication when pain remained bothersome.
  Additional analgesics may include primary analgesics (paracetamol and/or opioids) and/or adjuvant analgesics (muscle relaxants, antiepileptics, antidepressants, antispasmodics).

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee of Faculty of Medicine
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No